CLINICAL TRIAL: NCT03903653
Title: Effects of Chemodenervation (Botulinum Toxin A) and Serial Casting vs Botulinum Toxin A and Without Serial Casting in Lower Limb Spasticity Following ABI
Brief Title: Botulinum Toxin A & Weekly Serial Casting in ABI Inpatients With Lower Extremity Spasticity
Acronym: ChemoCast
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll patients due to closure of our inpatient units secondary to COVID-19.
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Ali Fateh, Resident - Dept of Physical Medicine and Rehabilitation, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5301
Record Dates: First submitted 2018-12-02; First posted 2019-04-04 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Spastic Foot
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemodenervation + Serial Casting (Active Comparator): in this group a total of 10 patients will undergo Botulinum Toxin A injection and weekly serial casting Intervention = Weekly Serial Casting AND Botulinum Toxin A injection (350-400 units per treated limb)
  Interventions: Drug: Botulinum toxin type A; Device: Serial Casting
- Chemodenervation without serial casting (Active Comparator): in this group a total of 10 patients will undergo Botulinum Toxin A injection. Intervention = Botulinum Toxin A injection (350-400 units per treated limb) alone.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Use of chemodenervation (botulinum toxin A) for treatment of lower extremity spasticity in ABI inpatients with regards to ankle range of motion.
  (a total of 350-400 units of botulinum toxin A per treated limb)
  Other Names: Botox
Device: Serial Casting — Using Serial Casting in conjunction with Botox injection for treatment of lower extremity spasticity in ABI inpatients with regards to ankle range of motion.
  (a total of 350-400 units of botulinum toxin A per treated limb)
  Other Names: Casting
  Arms: Chemodenervation + Serial Casting

SUMMARY:
Effects of Chemodenervation (Botulinum Toxin A) and Serial Casting vs Botulinum Toxin A and without serial casting in Lower Limb Spasticity following ABI.

DETAILED DESCRIPTION:
The investigators will be studying the effects of Chemodenervation (Botulinum Toxin A) and Serial Casting vs Botulinum Toxin A and without serial casting in Lower Limb Spasticity following ABI.

patients are randomly divided into two groups: group 1 will undergo botox injection with weekly serial casting group 2 will undergo botox injection with physiotherapy The primary outcome is the effects of the proposed treatment with respect to passive dorsiflexion.

ELIGIBILITY:
Inclusion Criteria

* Patients with Acquired Brain Injury (ABI) including but not limited to stroke, traumatic and anoxic brain injury in ABI unit of RRC
* Dorsiflexion limitation of < 10 degrees from neutral and Modified Ashworth Score (MAS) of 2 or 3
* Patients that are on Oral Medication for Spasticity Tx are still allowed to participate (ie. Baclofen)
* Patients both with Bilateral or Unilateral Lower Limb Spasticity are included
* There will be no sex or age restrictions

Exclusion Criteria

* Patients cannot have had Botulinum Toxin A Injections in their Lower Extremities within the past 6 months
* Patients cannot have had any sort of custom bracing or serial casting previously
* Patients with MAS of 4
* Patients with generalized spasticity that require other alternative treatment such as intra-thecal baclofen or surgical intervention
* Patients need to be medically stable (all co-morbidities under control via medical/pharmacological therapy), patients with ongoing co-morbid medical condition that are unmanaged will be excluded.
* Patients whom have skin breakdown in their lower extremities prior to the study will be excluded
* Patients who develop Skin breakdown (Grade 2 or higher) during the course of the study will be removed automatically

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Passive ankle dorsiflexion >10 degrees | 4-6 weeks
  we are measuring passive ankle range of motion with respect to dorsiflexion greater than 10 degrees

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Hossein Hosseini, M.D., Principal Investigator — Hamilton Health Sciences Corporation

IPD SHARING:
Plan to Share IPD: Undecided